CLINICAL TRIAL: NCT07358793
Title: Effectiveness of In Situ and Off-site Simulation on A-C-L-S Teamwork Model Implementation for Adult Non-trauma Resuscitation: A Two-group Pre-post Study
Brief Title: Effectiveness of In-Situ Simulation Training in Adult Non-Trauma Resuscitation: A Comparison of ISS and OSS Team Performance Using the A-C-L-S Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202510146RIND
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Adult Non-trauma Cardiac Arrest Resuscitation; Effectiveness of In-situ Simulation (ISS) Training; Effectiveness of Off-site Simulation (OSS) Training; Improvement of Teamwork in Emergency Care Settings
Keywords: In-situ Simulation; Teamwork; Resuscitation; Interprofessional Training; TEAM Scale

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-situ Simulation (ISS) Group (Experimental)
  Interventions: Other: In-situ Simulation (ISS) Training
- Off-site Simulation (OSS) Group (Active Comparator)
  Interventions: Other: Off-site Simulation (OSS) Training

INTERVENTIONS:
Other: In-situ Simulation (ISS) Training — The ISS group will undergo high-fidelity simulation training conducted in a real clinical environment, such as the emergency department. This training will involve a structured scenario with a briefing (20 minutes), a simulation exercise (10 minutes), and a debriefing session (30 minutes). The goal is to enhance teamwork and improve non-technical skills (e.g., communication, coordination) during adult non-trauma cardiac arrest resuscitation. The training follows the A-C-L-S (Airway-Circulation-Leadership-Support) model for team role structuring.
  Arms: In-situ Simulation (ISS) Group
Other: Off-site Simulation (OSS) Training — The OSS group will participate in simulation training at a dedicated simulation center, using high-fidelity mannequins and equipment. Similar to the ISS group, the training involves a briefing (20 minutes), a simulation scenario (10 minutes), and a debriefing (30 minutes). However, this training is conducted in a controlled environment away from the real clinical setting. The training follows the same A-C-L-S model for team role structuring and focuses on improving teamwork and technical skills for resuscitation.
  Arms: Off-site Simulation (OSS) Group

SUMMARY:
This study employed a two-group non-randomized pre-post design to evaluate the effectiveness of interprofessional ISS training over one year at the National Taiwan University Hospital Yunlin Branch. The research implements the A-C-L-S teamwork model for adult non-trauma resuscitation teams, comparing the impacts of ISS versus Off-site Simulation (OSS) on team performance. Emergency department teams are assigned between two campuses: ISS at Douliu campus and OSS at Huwei campus. Each training session follows a standardized protocol: twenty-minute briefing, ten-minute high-fidelity simulation, and thirty-minute structured debriefing. The assessment utilizes the Team Emergency Assessment Measure (TEAM) scale for non-technical skills evaluation, alongside secondary outcomes including resuscitation process, CPR quality, and patient outcome indicators. External ACLS instructor-qualified experts conduct blinded evaluations of recorded scenarios to analyze team performance and training transfer. The study aims to deliver benefits across three dimensions: establishing evidence-based education models to enhance resuscitation team efficiency and patient outcomes; strengthening institutional teaching and research capacity through standardized assessment mechanisms; and developing systematic data collection processes with localized quality indicators for early error detection and improvement.

ELIGIBILITY:
Inclusion Criteria:

The Adult Non-Traumatic Resuscitation Teams in the emergency departments of the Douliu and Huwei (branches consist of approximately 2 to 7 healthcare professionals per team). The healthcare professionals include attending physicians, resident physicians, specialized nurses, and registered nurses from the National Taiwan University Hospital system.

Exclusion Criteria:

1. Medical students and emergency medical technicians (EMTs) observing resuscitation in the emergency room.
2. Healthcare professionals who have not obtained a valid ACLS certification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Non-Technical Skills Evaluation Using the TEAM Scale | Through study completion, an average of 1 year
  The Team Emergency Assessment Measure (TEAM) scale will be used to evaluate non-technical skills. The scale consists of 11 items across three categories (leadership, teamwork, and task management) and a global rating. Total scores range from 0 to 44, where higher scores represent better team performance and non-technical skills.

SECONDARY OUTCOMES:
Time to Key Resuscitation Interventions | Through study completion, an average of 1 year.
  This measure assesses the efficiency of the ACLS team. We will measure the time intervals (in seconds/minutes) for critical steps, including:
  1. Time to initial pulse and rhythm assessment.
  2. Time to first shock (for shockable rhythm).
  3. Time to first adrenaline (for non-shockable rhythm).
  4. Time to endotracheal intubation completion.
  5. Time to established EtCO2 monitoring.
  6. Time to first ultrasound exam.
CPR Quality - Chest Compression Fraction (CCF) | Through study completion, an average of 1 year.
  The Chest Compression Fraction (CCF) is defined as the proportion of total resuscitation time during which active chest compressions are performed. It is calculated by dividing the total chest compression time by the total duration of the resuscitation event. This indicator is used to evaluate the resuscitation team's ability to minimize interruptions during cardiopulmonary resuscitation (CPR). Data will be collected through systematic observation and analysis of resuscitation performance during both in-situ and off-site simulation training, as well as actual clinical events, to assess the effectiveness of the A-C-L-S teamwork model.
Patient Outcomes - Rate of Return of Spontaneous Circulation (ROSC) | Through study completion, an average of 1 year.
  The percentage of patients achieving Return of Spontaneous Circulation (ROSC) after cardiac arrest. ROSC is defined as the restoration of a palpable pulse and measurable blood pressure during the resuscitation process. This measure evaluates the clinical outcome of the A-C-L-S teamwork model. Data collection includes comprehensive analysis of patient outcomes and factors influencing resuscitation success, such as initial cardiac rhythm, cause of arrest, and pre-hospital interventions, to assess the overall effectiveness of the simulation training.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch (Douliu), Douliu, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mei Q, Zhang T, Chai J, Liu A, Liu Y, Zhu H. Application of In Situ Scenario Simulation in Advanced Cardiac Life Support Training for Eight-year Medicinal Students. Medical Journal of Peking Union Medical College Hospital. 2023;14(3):660-664. doi:10.12290/xhyxzz.2022-0676
- [Background] Cooper S, Cant R, Connell C, Sims L, Porter JE, Symmons M, Nestel D, Liaw SY. Measuring teamwork performance: Validity testing of the Team Emergency Assessment Measure (TEAM) with clinical resuscitation teams. Resuscitation. 2016 Apr;101:97-101. doi: 10.1016/j.resuscitation.2016.01.026. Epub 2016 Feb 11. PMID 26875992
- [Background] Maignan M, Koch FX, Chaix J, Phellouzat P, Binauld G, Collomb Muret R, Cooper SJ, Labarere J, Danel V, Viglino D, Debaty G. Team Emergency Assessment Measure (TEAM) for the assessment of non-technical skills during resuscitation: Validation of the French version. Resuscitation. 2016 Apr;101:115-20. doi: 10.1016/j.resuscitation.2015.11.024. Epub 2015 Dec 17. PMID 26708450
- [Background] Cooper S, Connell C, Cant R. Review article: Use of the Team Emergency Assessment Measure in the rating of emergency teams' non-technical skills: A mapping review. Emerg Med Australas. 2023 Jun;35(3):375-383. doi: 10.1111/1742-6723.14184. Epub 2023 Feb 27. PMID 36849717
- [Background] Smidt A, Balandin S, Sigafoos J, Reed VA. The Kirkpatrick model: A useful tool for evaluating training outcomes. J Intellect Dev Disabil. 2009 Sep;34(3):266-74. doi: 10.1080/13668250903093125. PMID 19681007
- [Background] Cortegiani A, Ippolito M, Abelairas-Gomez C, Nabecker S, Olaussen A, Lauridsen KG, Lin Y, Sawyer T, Yeung J, Lockey AS, Cheng A, Greif R; International Liaison Committee on Resuscitation Education, Implementation and Teams Task Force (EIT) Task Force. In situ simulation for cardiopulmonary resuscitation training: A systematic review. Resusc Plus. 2025 Jan 3;21:100863. doi: 10.1016/j.resplu.2024.100863. eCollection 2025 Jan. PMID 39897060
- [Background] Riley W, Davis S, Miller K, Hansen H, Sainfort F, Sweet R. Didactic and simulation nontechnical skills team training to improve perinatal patient outcomes in a community hospital. Jt Comm J Qual Patient Saf. 2011 Aug;37(8):357-64. doi: 10.1016/s1553-7250(11)37046-8. PMID 21874971
- [Background] Hunt EA, Hohenhaus SM, Luo X, Frush KS. Simulation of pediatric trauma stabilization in 35 North Carolina emergency departments: identification of targets for performance improvement. Pediatrics. 2006 Mar;117(3):641-8. doi: 10.1542/peds.2004-2702. PMID 16510642
- [Background] Hunt EA, Heine M, Hohenhaus SM, Luo X, Frush KS. Simulated pediatric trauma team management: assessment of an educational intervention. Pediatr Emerg Care. 2007 Nov;23(11):796-804. doi: 10.1097/PEC.0b013e31815a0653. PMID 18007210
- [Background] Steinemann S, Berg B, Skinner A, DiTulio A, Anzelon K, Terada K, Oliver C, Ho HC, Speck C. In situ, multidisciplinary, simulation-based teamwork training improves early trauma care. J Surg Educ. 2011 Nov-Dec;68(6):472-7. doi: 10.1016/j.jsurg.2011.05.009. Epub 2011 Aug 3. PMID 22000533
- [Background] Carayon P, Schoofs Hundt A, Karsh BT, Gurses AP, Alvarado CJ, Smith M, Flatley Brennan P. Work system design for patient safety: the SEIPS model. Qual Saf Health Care. 2006 Dec;15 Suppl 1(Suppl 1):i50-8. doi: 10.1136/qshc.2005.015842. PMID 17142610
- [Background] Weaver SJ, Rosen MA, Salas E, Baum KD, King HB. Integrating the science of team training: guidelines for continuing education. J Contin Educ Health Prof. 2010 Fall;30(4):208-20. doi: 10.1002/chp.20085. PMID 21171026
- [Background] Zendejas B, Cook DA, Bingener J, Huebner M, Dunn WF, Sarr MG, Farley DR. Simulation-based mastery learning improves patient outcomes in laparoscopic inguinal hernia repair: a randomized controlled trial. Ann Surg. 2011 Sep;254(3):502-9; discussion 509-11. doi: 10.1097/SLA.0b013e31822c6994. PMID 21865947
- [Background] Issenberg SB, McGaghie WC, Hart IR, Mayer JW, Felner JM, Petrusa ER, Waugh RA, Brown DD, Safford RR, Gessner IH, Gordon DL, Ewy GA. Simulation technology for health care professional skills training and assessment. JAMA. 1999 Sep 1;282(9):861-6. doi: 10.1001/jama.282.9.861. PMID 10478693
- [Background] Merien AER, van de Ven J, Mol BW, Houterman S, Oei SG. Multidisciplinary team training in a simulation setting for acute obstetric emergencies: a systematic review. Obstet Gynecol. 2010 May;115(5):1021-1031. doi: 10.1097/AOG.0b013e3181d9f4cd. PMID 20410778
- [Background] Weaver SJ, Salas E, Lyons R, Lazzara EH, Rosen MA, Diazgranados D, Grim JG, Augenstein JS, Birnbach DJ, King H. Simulation-based team training at the sharp end: A qualitative study of simulation-based team training design, implementation, and evaluation in healthcare. J Emerg Trauma Shock. 2010 Oct;3(4):369-77. doi: 10.4103/0974-2700.70754. PMID 21063560
- [Background] Eppich W, Howard V, Vozenilek J, Curran I. Simulation-based team training in healthcare. Simul Healthc. 2011 Aug;6 Suppl:S14-9. doi: 10.1097/SIH.0b013e318229f550. PMID 21817858
- [Background] Issenberg SB, McGaghie WC, Petrusa ER, Lee Gordon D, Scalese RJ. Features and uses of high-fidelity medical simulations that lead to effective learning: a BEME systematic review. Med Teach. 2005 Jan;27(1):10-28. doi: 10.1080/01421590500046924. PMID 16147767
- [Background] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Background] Chong KM, Chou EH, Chiang WC, Wang HC, Liu YP, Ko PC, Huang EP, Hsieh MJ, Lin HY, Lien WC, Huang CH, Fang CC, Chen SC, Bhanji F, Yang CW, Ma MH. Development and Evaluation of a Novel Resuscitation Teamwork Model for Out-of-Hospital Cardiac Arrest in the Emergency Department. Ann Emerg Med. 2025 Feb;85(2):163-178. doi: 10.1016/j.annemergmed.2024.09.008. Epub 2024 Nov 8. PMID 39520453
- [Background] Aitken M, Gorokhovich L. Advancing the Responsible Use of Medicines: Applying Levers for Change. SSRN Electronic Journal. Sep 17 2012;doi:10.2139/ssrn.2222541
- [Background] Panagioti M, Khan K, Keers RN, Abuzour A, Phipps D, Kontopantelis E, Bower P, Campbell S, Haneef R, Avery AJ, Ashcroft DM. Prevalence, severity, and nature of preventable patient harm across medical care settings: systematic review and meta-analysis. BMJ. 2019 Jul 17;366:l4185. doi: 10.1136/bmj.l4185. PMID 31315828
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Care Services; Board on Global Health; Committee on Improving the Quality of Health Care Globally. Crossing the Global Quality Chasm: Improving Health Care Worldwide. Washington (DC): National Academies Press (US); 2018 Aug 28. Available from http://www.ncbi.nlm.nih.gov/books/NBK535653/ PMID 30605296
- See also: Related Info — https://cpredu.com/knowledge-base/resuscitation-triangle-roles-in-a-high-performance-team/